CLINICAL TRIAL: NCT01145612
Title: A Clinical Trial to Assess the Efficacy and Safety of Losartan Versus Atenolol in the Prevention of Progressive Dilation of the Aorta in Patients With Marfan Syndrome.
Brief Title: Atenolol Versus Losartan in the Prevention of Progressive Dilation of the Aorta in Marfan Syndrome
Acronym: LO-AT-MARFAN01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Forteza, Albert, M.D. (Individual)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Dr Alberto Forteza, Dr Alberto Forteza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LO-AT-MARFAN-01; 2007-001125-97 (EudraCT Number)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-06

CONDITIONS: Marfan Syndrome
Keywords: Aortic dilation; Marfan syndrome; Losartan; Atenolol
MeSH Terms: conditions — Marfan Syndrome | interventions — Losartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Experimental): Losartán dosage: 12.5 mg /day for patients < 50 Kg or 25 mg/day for patients > 50 Kg (14 days). 50 mg/day from day 15 to the end of the study. Half of dose (25 mg/day) for patients < 50 Kg
  Interventions: Drug: Losartan
- Atenolol (Experimental): Atenolol dosage: 12.5 mg /day for patients < 50 Kg or 25 mg/day for patients > 50 Kg (14 days). 50 mg/day from day 15 to the end of the study. Half of dose (25 mg/day) for patients < 50 Kg
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Losartan — Losartán dosage: 12.5 mg /day for patients < 50 Kg or 25 mg/day for patients > 50 Kg (14 days). 50 mg/day from day 15 to the end of the study. Half of dose (25 mg/day) for patients < 50 Kg
  Arms: Losartan
Drug: Atenolol — Atenolol dosage: 12.5 mg /day for patients < 50 Kg or 25 mg/day for patients > 50 Kg (14 days). 50 mg/day from day 15 to the end of the study. Half of dose (25 mg/day) for patients < 50 Kg
  Arms: Atenolol

SUMMARY:
The purpose of this study is to evaluate the efficacy of Losartan versus Atenolol in the progression of aortic dilatation in patients with Marfan syndrome.

DETAILED DESCRIPTION:
Marfan syndrome is a genetic disease of the connective tissue. Patients with Marfan syndrome experience an expansion of the aorta that can lead to dissection or rupture of it. This is the main cause of mortality in these patients.

The main objective of this study is to evaluate the efficacy of Losartan versus Atenolol in the progression of aortic dilation in patients with Marfan syndrome.

The measurement is made by echocardiography, assessing the diameter of the aorta in different zones: valve annulus, sinuses of Valsalva, sinotubular junction, ascending aorta, aortic arch, thoracic and abdominal aorta.

A total number of 150 subjects diagnosed with Marfan syndrome and who meet the diagnostic criteria of Ghent, of both sexes, 75 per treatment group, aged between 5 and 60, will be included in the study. The study is being conducted in two Spanish hospitals.

The treatment is maintained throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must conform to the diagnostic criteria Marfan syndrome according to the Ghent Criteria.
2. Outpatient subjects.
3. Male or female, aged between 5 and 60 years.
4. Women who are in a childbearing age are required a result of negative Gonadotropin pregnancy test to be included in the study.
5. Subjects must be able to take oral medication.
6. After having received information about the study, subjects must understand the nature of it and give written informed consent.
7. For Subjects under 18 years, the informed consent must be signed by their parents or guardians.
8. Subjects with a maximum diameter of the aorta, at length, <45 mm
9. Female subjects of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for four weeks prior to, during and three months after the last dose study medication.

For the purposes of this study, women of childbearing potential is defined as: All female subjects after puberty unless they are post-menopausal for at least two years, or are surgically sterile. Adequate contraception is defined as two barrier methods, or one barrier method with a spermicide, or an intrauterine device or use of the oral female contraceptive (or other hormonal methods).

Exclusion Criteria:

1. Women who are pregnant, suspected to be pregnant or breast-feeding.
2. Ongoing participation in another clinical trial or who received the investigational drug in the month prior to the inclusion in the study.
3. Known or suspected failure to comply with the study protocol.
4. Previous surgery: cardiac or at any segment of the aorta.
5. Functional class III-IV.
6. Maximum diameter of the aorta exceeding 45 mm
7. More than moderate valvular involvement.
8. History or presence of respiratory failure, liver (ALT> 3 x ULN), renal (creatinine clearance <30 mL / min), gastrointestinal, hematological, endocrine, or any other situation that may affect the assessment of the study treatment, according to the investigator opinion.
9. History of aortic dissection.
10. History or presence of neurological disease (especially seizures, dementia ...).
11. History or presence of alcohol abuse and / or toxic substances
12. Uncontrolled depression.
13. Any need for another antihypertensive treatment (betablockers, diuretics, calcium channel blockers, ACE inhibitors, ARBs, etc.)
14. Hypersensitivity, intolerance or contraindication to any component of the study drug.
15. Patients with a history of drug abuse or toxic dependence.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2008-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Progression of aortic dilation in patients with Marfan syndrome. | Until February 2013
  Evaluate the eficacy of Losartan versus Atenolol in the progression of aortic dilation in patients with Marfan syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Forteza, Dr, Principal Investigator; Arturo Evangelista, Dr, Principal Investigator
Locations (2):
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid, Madrid